CLINICAL TRIAL: NCT05999188
Title: Clinical Characteristics and Prognosis of Aortic Dissection in China (CLASSIC): a National, Multicenter, Retrospective-prospective, Cohort Study
Brief Title: Clinical Characteristics and Prognosis of Aortic Dissection in China (CLASSIC)
Acronym: CLASSIC
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Collaborators: 521 Hospital of NORINCO Group (Other); Shaanxi Provincial People's Hospital (Other); Xiangyang Central Hospital (Other); Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF2023LSK-313
Record Dates: First submitted 2023-08-13; First posted 2023-08-21 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-04

CONDITIONS: Aortic Dissection
Keywords: aortic dissection; clinical characteristics; prognosis
MeSH Terms: conditions — Aortic Dissection | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Blood, urine, faeces, other types of body fluids (e.g. pericardial fluid), surgical and biopsy collected tissue specimens.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aortic dissection group: Patients diagnosed with aortic dissection at any of the centres and regularly consulted and followed up.
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — No interventions will be given to patients.

SUMMARY:
This study will construct a retrospective-prospective long-term follow-up cohort and management system for aortic dissection through a multicentre collaborative network. This study aims to investigate the disease characteristics, progression patterns, clinical features, natural course and factors affecting the disease course and prognosis of patients with aortic dissection by retrospectively collecting data and prospectively enrolling patients.

DETAILED DESCRIPTION:
This study aims to construct a retrospective-prospective long-term follow-up cohort and management system for aortic dissection through a multicentre collaborative network. The duration of the study will be divided into retrospective and prospective components. The retrospective study will collect cases of aortic dissection of different aetiologies from 2003-2022; the prospective study is expected to collect cases of aortic dissection from 2022-2030. The study is expected to assess the disease characteristics, progression patterns, clinical features, natural course and long-term prognosis of aortic coarctation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years;
* Meet diagnostic criteria for aortic dissection.

Exclusion Criteria:

* Age <18 years or >80 years;
* Women who are pregnant and breastfeeding;
* Patients and their families refuse or are unable to sign the informed consent form.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are aged 18-80 years and diagnosed with aortic dissection at any of the centre can be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2030-10-12 (Estimated); Study Completion 2030-12-12 (Estimated)

PRIMARY OUTCOMES:
Change of post-operative survival rate | 3, 6, 9 month and 1, 2, 3, 4, 5 year after the surgery.
  Post-operative survival rate of patients after aortic dissection surgery in 3, 6, 9 month and 1, 2, 3, 4, 5 year. The survival situation will be assessed by telephone follow-up.

SECONDARY OUTCOMES:
Change of the incidence of MACCE | 3, 6, 9 month and 1, 2, 3, 4, 5 year after the surgery.
  Major adverse cardio-cerebrovascular events included myocardial infarction, stroke, revascularization and all-cause death. The occurrence of MACCE will be assessed by telephone follow-up and medical records.
Incidence of any complications | 5 years after the surgery.
  Any complications diagnosed by doctors. The occurrence of complications will be decided by medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Guoliang Li, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University; Yang Yan, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xian Jiantong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No